CLINICAL TRIAL: NCT03828786
Title: The Impact of Uterine Scratching Prior to Intra-Uterine Insemination in Unexplained Infertility, a Randomized Controlled Trial
Brief Title: Uterine Scratching in Intra-Uterine Insemination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ovo-18-01
Record Dates: First submitted 2018-07-27; First posted 2019-02-04 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Infertility; Unexplained Infertility
Keywords: intra-uterine insemination; endometrial injury; scratching
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endometrial scratching group (Active Comparator): Endometrial scratching will be done with a Pipelle in uterus.
  Interventions: Procedure: Endometrial scratching
- Control group (No Intervention): This group will proceed with intrauterine insemination without endometrial scratching according to clinic's standard procedure

INTERVENTIONS:
Procedure: Endometrial scratching — Endometrial Biopsy by aspiration with a pipelle
  Other Names: Endometrial Biopsy
  Arms: Endometrial scratching group

SUMMARY:
This study will evaluate the potential benefits of uterine injury during the follicular phase of an intra-uterine insemination cycle on the rate of ongoing pregnancy during the first trimester ultrasound.

DETAILED DESCRIPTION:
Infertility is defined as the absence of conception after a year of unprotected intercourse. In 10 to 30 % of patients, the cause of the infertility is unknown. An emerging practice in unexplained infertility has been to cause a uterine trauma prior to treatment. This is done by doing a small endometrial scratch with a pipelle. This intervention has been study in IVF and has been shown beneficial. Theoretically, the uterine scratching could increase the immune response and the vascularization of the endometrium which could help in embryo implantation. However, there is very few data concerning scratching in intrauterine insemination. The studies are mostly small studies and the results are often contradictory. In this randomized controlled trial, the investigators will evaluate the effect of uterine scratching during the follicular phase of an insemination cycle on the pregnancy rate of a large cohort of unexplained infertile couples.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained infertility for over 12 months if under 35 years old or over 6 months if 35 years old and above.
* At least one permeable tube on hysterosonography or hysterosalpingography within the last 2 years or vaginal delivery in the last 3 years.
* Antral follicular count over 5.
* Normal or mild male factor.
* Normal uterine cavity.
* An IUI prescription.

Exclusion Criteria:

* Polycystic ovary syndrome with irregular menstrual cycles over 45 days
* Severe endometriosis
* IUI with Donor sperm
* Patient with invasive intra-uterine procedure in the last 3 months.
* Contraindication to endometrial biopsy.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women of reproductive age
Enrollment: 394 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Efficacy - Pregnancy Rate measured during the first trimester ultrasound. | 13 weeks
  Ongoing pregnancy during the first trimester ultrasound after an intrauterine insemination (IUI) cycle.

SECONDARY OUTCOMES:
Efficacy - Secondary pregnancy rate. | 6 months
  Ongoing pregnancy during the first trimester ultrasound in the 3 IUI cycles following a scratching
Safety - Side effects | 6 months for all 3 intrauterine insemination
  Evaluate side effects related to the intrauterine scratching
Safety - Complications | 6 months for all 3 intrauterine insemination
  Evaluate complications related to intrauterine scratching

CONTACTS AND LOCATIONS:
Overall Officials: Louise Lapensee, Md, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou L, Li R, Wang R, Huang HX, Zhong K. Local injury to the endometrium in controlled ovarian hyperstimulation cycles improves implantation rates. Fertil Steril. 2008 May;89(5):1166-1176. doi: 10.1016/j.fertnstert.2007.05.064. Epub 2007 Aug 6. PMID 17681303
- [Background] Wadhwa L, Pritam A, Gupta T, Gupta S, Arora S, Chandoke R. Effect of endometrial biopsy on intrauterine insemination outcome in controlled ovarian stimulation cycle. J Hum Reprod Sci. 2015 Jul-Sep;8(3):151-8. doi: 10.4103/0974-1208.165144. PMID 26538858
- [Background] Raziel A, Schachter M, Strassburger D, Bern O, Ron-El R, Friedler S. Favorable influence of local injury to the endometrium in intracytoplasmic sperm injection patients with high-order implantation failure. Fertil Steril. 2007 Jan;87(1):198-201. doi: 10.1016/j.fertnstert.2006.05.062. PMID 17197286
- [Background] Practice Committee of the American Society for Reproductive Medicine. Definitions of infertility and recurrent pregnancy loss: a committee opinion. Fertil Steril. 2013 Jan;99(1):63. doi: 10.1016/j.fertnstert.2012.09.023. Epub 2012 Oct 22. PMID 23095139
- [Background] Nastri CO, Gibreel A, Raine-Fenning N, Maheshwari A, Ferriani RA, Bhattacharya S, Martins WP. Endometrial injury in women undergoing assisted reproductive techniques. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD009517. doi: 10.1002/14651858.CD009517.pub2. PMID 22786529
- [Background] Narvekar SA, Gupta N, Shetty N, Kottur A, Srinivas M, Rao KA. Does local endometrial injury in the nontransfer cycle improve the IVF-ET outcome in the subsequent cycle in patients with previous unsuccessful IVF? A randomized controlled pilot study. J Hum Reprod Sci. 2010 Jan;3(1):15-9. doi: 10.4103/0974-1208.63116. PMID 20607003
- [Background] Maged AM, Al-Inany H, Salama KM, Souidan II, Abo Ragab HM, Elnassery N. Endometrial Scratch Injury Induces Higher Pregnancy Rate for Women With Unexplained Infertility Undergoing IUI With Ovarian Stimulation: A Randomized Controlled Trial. Reprod Sci. 2016 Feb;23(2):239-43. doi: 10.1177/1933719115602776. Epub 2015 Sep 3. PMID 26342054
- [Background] Lensen SF, Manders M, Nastri CO, Gibreel A, Martins WP, Templer GE, Farquhar C. Endometrial injury for pregnancy following sexual intercourse or intrauterine insemination. Cochrane Database Syst Rev. 2016 Jun 14;(6):CD011424. doi: 10.1002/14651858.CD011424.pub2. PMID 27296541
- [Background] Lensen S, Sadler L, Farquhar C. Endometrial scratching for subfertility: everyone's doing it. Hum Reprod. 2016 Jun;31(6):1241-4. doi: 10.1093/humrep/dew053. Epub 2016 Mar 22. PMID 27008891
- [Background] Ledee N, Petitbarat M, Chevrier L, Vitoux D, Vezmar K, Rahmati M, Dubanchet S, Gahery H, Bensussan A, Chaouat G. The Uterine Immune Profile May Help Women With Repeated Unexplained Embryo Implantation Failure After In Vitro Fertilization. Am J Reprod Immunol. 2016 Mar;75(3):388-401. doi: 10.1111/aji.12483. Epub 2016 Jan 18. PMID 26777262
- [Background] Karimzadeh MA, Ayazi Rozbahani M, Tabibnejad N. Endometrial local injury improves the pregnancy rate among recurrent implantation failure patients undergoing in vitro fertilisation/intra cytoplasmic sperm injection: a randomised clinical trial. Aust N Z J Obstet Gynaecol. 2009 Dec;49(6):677-80. doi: 10.1111/j.1479-828X.2009.01076.x. PMID 20070722
- [Background] Gibreel A, Badawy A, El-Refai W, El-Adawi N. Endometrial scratching to improve pregnancy rate in couples with unexplained subfertility: a randomized controlled trial. J Obstet Gynaecol Res. 2013 Mar;39(3):680-4. doi: 10.1111/j.1447-0756.2012.02016.x. Epub 2012 Oct 29. PMID 23106834
- [Background] Finn CA, Martin L. Endocrine control of the timing of endometrial sensitivity to a decidual stimulus. Biol Reprod. 1972 Aug;7(1):82-6. doi: 10.1093/biolreprod/7.1.82. No abstract available. PMID 5050152
- [Background] Barash A, Dekel N, Fieldust S, Segal I, Schechtman E, Granot I. Local injury to the endometrium doubles the incidence of successful pregnancies in patients undergoing in vitro fertilization. Fertil Steril. 2003 Jun;79(6):1317-22. doi: 10.1016/s0015-0282(03)00345-5. PMID 12798877
- [Background] Bahaa Eldin AM, Abdelmaabud KH, Laban M, Hassanin AS, Tharwat AA, Aly TR, Elbohoty AE, Elsayed HM, Ibrahim AM, Ibrahim ME, Sabaa HM, Abdelrazik AA, Abdelhady I. Endometrial Injury May Increase the Pregnancy Rate in Patients Undergoing Intrauterine Insemination: An Interventional Randomized Clinical Trial. Reprod Sci. 2016 Oct;23(10):1326-31. doi: 10.1177/1933719116638191. Epub 2016 May 4. PMID 27146582
- [Background] Abdelhamid AM. The success rate of pregnancy in IUI cycles following endometrial sampling. A randomized controlled study: endometrial sampling and pregnancy rates. Arch Gynecol Obstet. 2013 Sep;288(3):673-8. doi: 10.1007/s00404-013-2785-0. Epub 2013 Mar 15. PMID 23494199